CLINICAL TRIAL: NCT00400530
Title: A Randomized, Single-Blind Study to Evaluate Upper Gastrointestinal Handling of Branded Versus Generic Alendronate Tablets
Brief Title: Upper GI Handling of Branded vs. Generic Alendronate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2006_050
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2006-11-17 (Estimated); Status verified 2006-11

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate; Duration of Therapy

INTERVENTIONS:
Drug: MK0217, alendronate sodium / Duration of Treatment: 1 Month
Drug: Comparator: Alendronate-Teva / Duration of Treatment: 1 Month

SUMMARY:
To compare upper GI handling of fosamax and generic, because the main AE profile of alendronate is before systemic absorption in the esophagus; differences could be relevant to the side effect profile.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal females aged greater 55 years
* Prescribed alendronate 70 mg tablets for a therapeutic indication throughout the previous 3 months and expected to continue on this treatment for the duration of the study
* Willing to abstain from alcohol for 24 hours before each dose and until the end of each study day
* Willing to abstain from smoking for 24 hours before each dose and until the end of each study day

Exclusion Criteria:

* History of drug hypersensitivity
* Suffers from dysphagia, achalasia, or other conditions or medications affecting upper gastrointestinal motility

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2005-12

PRIMARY OUTCOMES:
Gamma camera imaging of tablet dissolution in oesophagus

SECONDARY OUTCOMES:
Gamma camera dissolution of tablets in stomach

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC